CLINICAL TRIAL: NCT02107495
Title: Evaluation of the Samsung LABGEO IVD-A20 CHF Test in a Point-of-Care Setting
Status: Terminated | Type: Observational
Why Stopped: Optimize calibration
Sponsor: Samsung Electronics (Industry)
Collaborators: Nexus DX (Industry)
Responsible Party: Sponsor
Other Study IDs: A20-01
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2015-02

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Retaining plasma specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CHF-confirmed subjects: Subjects 21 years of age or greater with clinically confirmed heart failure or have presented to the clinical site with signs, symptoms and/or risk factors suggestive of heart failure.
  Interventions: Device: Samsung LABGEO IVD-A20 CHF Test
- Subjects with potentially co-morbidities: non-CHF subjects 21 years or greater, with potentially confounding comorbidities such as diabetes, renal insufficiency, hypertension and chronic obstructive pulmonary disease (COPD).
  Interventions: Device: Samsung LABGEO IVD-A20 CHF Test
- Apparently healthy subjects: Apparently healthy subjects (meeting inclusion criteria) greater than 45 years of age, with no prior history of myocardial infarction (MI), acute coronary syndrome (ACS) congestive heart failure (CHF) or any other cardiac-related disease.
  Interventions: Device: Samsung LABGEO IVD-A20 CHF Test

INTERVENTIONS:
Device: Samsung LABGEO IVD-A20 CHF Test
  Other Names: LABGEO IVD-A20 CHF Test, A20 CHF Test,

SUMMARY:
To establish the performance characteristics of the Samsung LABGEO IVD-A20 CHF Test in intended use settings, by comparing test results of the A20 CHF Test with results obtained from an FDA-cleared comparator assay.

ELIGIBILITY:
Inclusion Criteria:

* CHF Subjects: 21 years of age or greater, with clinically confirmed CHF or have presented to the clinical site with signs, symptoms and/or risk factors suggestive of heart failure.
* Subjects with Potentially confounding comorbidities: Non-CHF subjects 21 years of age or greater, with potentially confounding comorbidities such as diabetes, renal insufficiency, hypertension and chronic obstructive pulmonary disease (COPD)
* Healthy Subjects: apparently healthy subjects greater than 45 years of age, with no prior history of cardiac-related disease.

Exclusion Criteria:

* Apparently healthy subjects with a history of MI, CHF or other cardiac-related disease;
* Subjects with acute decompensated heart failure currently on nesiritide therapy;
* Subjects having participated in another experimental drug, biologic, or invasive device study within 30 days prior to signing informed consent for this study, or enrolled concurrently in any other investigative study; and
* Subjects unable to or refusing to provide written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects to be recruited for this study will be presenting to one of five point of care sites located in the USA. The sites will be emergency room or POL sites, and will include primary care facilities representative of those typically serving the intended use population for the test.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The proportion of clinically-confirmed CHF subjects for whom the Samsung LABGEO IVD-A20 CHF Test result was positive (clinical sensitivity). | baseline
The proportion of non-CHF subjects for whom the LABGEO IVD A20 CHF Test result was negative (clinical specificity). | baseline
Using a Passing-Bablok regression analysis, estimates of intercept and slope will be computed. Estimates of bias and corresponding 95% confidence interval for true bias at clinical decision threshold of 125mg/mL and 450 pg/mL will also be computed. | baseline
  Method comparison will be assessed using a Passing-Bablok regression analysis to determine the relationship between the Samsung LABGEO IVD-A20 CHF Test measurement in plasma and the corresponding measurement in plasma obtained from the comparator assay.

SECONDARY OUTCOMES:
The proportion of subjects with a positive LABGEO IVD-A20 CHF Test result, for whom a clinical diagnosis of CHF was confirmed (positive predictive value). | baseline
The proportion of subjects with a negative LABGEO IVD-A20 CHF Test result, for whom a clinical diagnosis of CHF was confirmed (negative predictive value). | baseline
Computation of Receiver Operating Characteristic (ROC) curve and area under the curve (AUC) with 95% confidence interval for the true AUC. | baseline
  This analysis will assess the ability of the Samsung LABGEO IVD-A20 CHF Test to discriminate between confirmed CHF subjects and non-CHF subjects.
Variance components analysis will be conducted on data collected from each whole blood specimen undergoing point-of-care precision testing at study site. Estimates of within-run, between run, between day and total precision will be computed. | 10 days
  The Samsung LABGEO IVD-A20 CHF Test result will be modeled as a function of testing days and runs, with replicates fully nested within runs, and runs fully nested within days.
Variance components analysis will be conducted on data collected from each plasma specimen undergoing point-of-care precision testing at study site. Estimates of within-run, between run, between day and total precision will be computed. | 20 days
  The Samsung LABGEO IVD-A20 CHF Test result will be modeled as a function of testing days and runs, with replicates fully nested within runs, and runs fully nested within days.
Mixed model regression analysis will be conducted on each specimen type (whole blood vs. plasma) and storage condition. | 48 hours
  The natural logarithm of the Samsung LABGEO IVD-A20 CHF Test measurement will be modeled as a linear function of time (in hours) after baseline testing.A separate linear function will be fitted to data collected from each study specimen and the intercepts and slops from individual specimens will be modeled as random effects.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Maryland
  - Minneapolis Medical Research Foundation, Minneapolis, Minnesota
  - Manassas Clinical Research Center, Manassas, Virginia